CLINICAL TRIAL: NCT03654144
Title: Role of Dienogest in the Treatment of Patient With Symptomatic Adenomyosis
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, asmaa mohamed hussin yousef, Principal investigator, Assiut University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DINADEN
Record Dates: First submitted 2018-08-29; First posted 2018-08-31 (Actual); Last update posted 2018-08-31 (Actual); Status verified 2018-08

CONDITIONS: Adenomyosis
MeSH Terms: conditions — Adenomyosis | interventions — dienogest; Contraceptives, Oral, Combined

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Study group (Experimental): women will receive dienogest
  Interventions: Drug: Dienogest
- control group (Active Comparator): women used combined oral contraceptive pills
  Interventions: Drug: Combined Oral Contraceptive

INTERVENTIONS:
Drug: Dienogest — oral tablets
  Arms: Study group
Drug: Combined Oral Contraceptive — oral tablets
  Arms: control group

SUMMARY:
Adenomyosis was first described as endometrial glands in the myometrium of the uterus. The current definition of adenomyosis is provided in 1972 'the benign invasion of endometrium into the myometrium, producing a diffusely enlarged uterus which microscopically exhibits ectopic non-neoplastic, endometrial glands and stroma surrounded by the hypertrophic and hyperplastic myometrium

ELIGIBILITY:
Inclusion Criteria:

* symptomatic adenomyosis
* irregular menstrual bleeding and dysmenorrhea .

Exclusion Criteria:

* asymptomatic patients -
* non-lactating patient
* not desire for pregnancy
* no hormonal treatment more than 6 month even contraception e.g IUD
* no focal lesion of uterus (malignancy ,fibroid or adenxal mass )

Min Age: 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2018-11 (Estimated); Primary Completion 2019-12 (Estimated); Study Completion 2020-03 (Estimated)

PRIMARY OUTCOMES:
The mean pain score after receiving treatment | 6 months
  assessment by visual analog scale